CLINICAL TRIAL: NCT04041024
Title: Identification of Decision Making Processes in Food, Risky and Steal Situations in Bulimia Nervosa
Brief Title: Decision-making and Risk-taking in Bulimia
Acronym: FaciB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI has left the hospital and no one is replacing him
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-A01268-47
Record Dates: First submitted 2019-07-25; First posted 2019-08-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Bulimia Nervosa
Keywords: computational psychiatry; decision making; risk; food; monetary; eating disorder
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bulimia nervosa group (Experimental): Patients with Bulimia Nervosa according to DSM 5 criteria aged between 18 and 35 years and specifically for participants attending MRI scans in the experiments: no counter indication to MRI scans and right handed.
  Interventions: Other: tasks and questionnaires
- Control group (Other): healthy participants without any history of eating disorder aged between 18 and 35 years and specifically for participants attending MRI scans in the experiments: no counter indication to MRI scans and right
  Interventions: Other: tasks and questionnaires

INTERVENTIONS:
Other: tasks and questionnaires — Each of the 4 experiments is built of a main task. The first task involves a first phase of subjective valuation of food items.
  The second phase requires from the participant to make a choice between two out of three food items selected by the computer.
  Arms: bulimia nervosa group
Other: tasks and questionnaires — Each of the 4 experiments is built of a main task. The first task involves a first phase of subjective valuation of food items.
  The second phase requires from the participant to make a choice between two out of three food items selected by the computer.
  Arms: Control group

SUMMARY:
This trial is a set of four independent experiments involving for each of them functional and structural MRI data acquisition. They aim at investigating decision making mechanisms in bulimia nervosa when participants have to make food or monetary choices under specific conditions that mimic binge eating episodes or kleptomania which are two major symptoms of bulimia nervosa. All experiments are cross sectional studies. Each experiment is subdivided into two parts: a first part without any MRI data acquisition and during which all the tasks are performed. This part aims at making sure that a behavioral effect is observed before starting MRI data acquisition. The second part aims at investigating the neural correlates observed in the first part and additionally, at reproducing the behavioral effects observed in the first part. Therefore the first part may be regarded as an independent study as compared to the second part.

DETAILED DESCRIPTION:
Each part of each experiment is built of a main task, a set of secondary tasks and questionnaires. Only the main task changes from one experiment to another. Within each experiment, the only difference between the two parts is that the main task is performed while participants are being scanned in an MRI scanner. Details of the tasks are provided below. Each part of each experiment is performed over one visit only and is a cross sectional study. The visit is dedicated to the tasks. Questionnaires may be filled during the visit or at participant's home within the week following the visit for questionnaires which are not assessing participant's state. Questionnaires assessing participant's state are filled during the visit at appropriate time. The total number of participants mentioned below is the sum of the planned number of participants within each group, i.e. patients and healthy participants, within each part of each experiment.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 18 to 35 years with bulimia nervosa according to DSM 5 criteria for the patient's group
* For the control group, men and women with the same age range being concerned by food intake and their body shape but without any history of eating disorder.
* All participants must have signed an informed consent form and be affiliated to the French public health insurance.
* for MRI scans, all participants must be right handed.

Exclusion Criteria:

* antisocial personality disorder,
* borderline personality disorder
* addiction to alcohol or psychoactive agent, ADHD, any psychotic disorder,
* obesity of class 1 or 2
* istory of psychiatric disorder for the control group
* history of neurological disorder for both groups
* intermittent explosive disorder
* any counter indication to MRI scans for the parts of experiments which take place in the MRI scanner.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
oxygen variation in the brain | 10 days
  Brain activity related to task performance collected in the MRI scanner.Blood Oxygen Level Dependent response synchronized with any event of interest during the task. Events of interests are:
  * Onset time of any visual stimulus
  * Onset time of any response of the participant.

SECONDARY OUTCOMES:
Task related parameters | 10 days
  reaction times computed as the duration in ms between the onset time of the stimulus and the onset time of the participant's answer. Several tasks may be involved in each experiment including in the MRI scan.
  These rules apply to all tasks.
Skin conductance response related to events in the task performed while the signal is being collected | 10 days
  Skin conductance response in microSiemens synchronized with any event of interest during the task. Events of interests are:
  * Onset time of any visual stimulus
  * Onset time of any response of the participant
cardiac frequency in beats per minute related to events in the task performed while the signal is being collected | 10 days
  cardiac frequency is computed from the pulse plethysmogram sensor signal while the participant is performing the task. Task during which this signal is collected may be one of the tasks performed in the scanner as well as tasks performed outside the scanner.
parameters of eye movements extracted from the eye tracking signal is being collected | 10 days
  The parameters computed are X and Y position of the eye by amplitude of variation of pupil size over a time window synchronized with events in the task
Eating Disorders Examination (EDE-Q) | 10 days
  The EDE is a semi-structured interview conducted by a trained clinician to assess the psychopathology associated with the diagnosis of an eating disorder. The EDE is rated through the use of four subscales (restraint, eating concern, weight concern, shape concern) and global score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Vinatier, Lyon, Auvergne-Rhône-Alpes, France